CLINICAL TRIAL: NCT02273011
Title: Combined Spinal-epidural Versus Spinal Analgesia for Elective Caesarean Section in the Postoperative Period
Status: Completed | Type: Observational
Sponsor: Prof. Dr. med. Daniel Reuter (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. med. Daniel Reuter, Vice Medical Director, Universitätsklinikum Hamburg-Eppendorf
Organization: Universitätsklinikum Hamburg-Eppendorf (Other)
Other Study IDs: CSEvsSSSA
Record Dates: First submitted 2014-01-15; First posted 2014-10-23 (Estimated); Last update posted 2014-10-23 (Estimated); Status verified 2014-10

CONDITIONS: Satisfaction; Pain
MeSH Terms: conditions — Personal Satisfaction; Pain | interventions — Cesarean Section

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- single shot spinal anesthesia: single shot spinal anesthesia for caesarean section was executed for anesthesia, oral analgesic medication was applicated for postoperative analgesia.
  Interventions: Procedure: caesarean section
- combuned spinal epidural anesthesia: combined spinal epidural anesthesia for caesarean section was executed for anesthesia, epidural and oral analgesic medication was applicated for postoperative analgesia.
  Interventions: Procedure: caesarean section

INTERVENTIONS:
Procedure: caesarean section — elective caesarean section under regional anesthesia

SUMMARY:
Combined spinal epidural (CSEA) and single shot spinal anesthesia (SSSA) are both well-established anesthetic methods for caesarean section. CSEA combines the advantages of spinal anesthesia for the surgery, and epidural anesthesia for postoperative pain management. The aim of this randomized trial was to compare analgesia and patient satisfaction with CSEA continuous epidural administration of local anesthetics versus SSSA with oral pain medication in the postoperative period.

DETAILED DESCRIPTION:
Combined spinal epidural (CSEA) and single shot spinal anesthesia (SSSA) are both well-established anesthetic methods for caesarean section. CSEA combines the advantages of spinal anesthesia for the surgery, and epidural anesthesia for postoperative pain management. However, it is more time-consuming, and adds potentially risks of both single techniques.

The aim of this randomized trial was to compare analgesia and patient satisfaction with CSEA continuous epidural administration of local anesthetics versus SSSA with oral pain medication in the postoperative period.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists-physical status: I or II
* elective caesarean section

Exclusion Criteria:

* age under eighteen
* maternal systemic diseases
* allergies against the drugs used
* systemic infection or local infection in the puncture area
* dysfunctional coagulation
* coagulation-inhibiting drugs

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: healthy parturients scheduled for elective caesarean section
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2007-03; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
patient's satisfaction | perioperative
  Standardised questionnaire assessing pain, discomfort, anxiety

SECONDARY OUTCOMES:
additional oral pain medication | perioperative
  Assessment of additionally requested oral pain medication
pain score | perioperative
  Standardised questionnaire assessing pain by using the visual analogue scale

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Reuter, Principal Investigator — Universitätsklinukum Hamburg-Eppendorf
Locations (1):
- Universitätsklinikum Hamburg-Eppendorf, Hamburg, Hamburg, Germany